CLINICAL TRIAL: NCT04350528
Title: Comparison of Sedation Using Pentobarbital or Chlorpromazine in Pediatric Non-invasive Imaging Procedure: A Before and After Study
Brief Title: Comparison of Chlorpromazine or Pentobarbital Premedications for Pediatric Imaging Procedures
Acronym: PREIMAPED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PREIMAPED (29BRC19.0309)
Record Dates: First submitted 2020-03-30; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-03

CONDITIONS: Children Sedation
Keywords: Sedation; Medical imaging; Children; Pentobarbital; Chlorpromazine; Efficacy; Safety
MeSH Terms: interventions — Chlorpromazine; Pentobarbital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chlorpromazine
  Interventions: Drug: Chlorpromazine or Pentobarbital
- Pentobarbital
  Interventions: Drug: Chlorpromazine or Pentobarbital

INTERVENTIONS:
Drug: Chlorpromazine or Pentobarbital — Sedation

SUMMARY:
Sedation is often required for pediatric medical imaging procedures to ensure compliance and quality images. Recommendations exist regarding pediatric sedation, but there are currently no guidelines regarding the choice of the sedative drug. We aim to compare the efficacy and adverse events of per os pentobarbital with intravenous chlorpromazine in children undergoing diagnostic imaging procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children
* Sedation for the purpose of imaging
* Sedation using chlorpromazine or pentobarbital

Exclusion Criteria:

* Refusal to participate

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing sedation for the purpose of imaging in the pediatric department of Brest hospital
Sampling Method: Non-Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Sedation success | During the procedure
  Imaging purpose is answered

SECONDARY OUTCOMES:
Induction time | During the procedure
  Length of time required after the administration to achieve adequate sedation
Hospitalization duration | Through procedure completion
  Length of time from planned time of admission to discharge
Duration of the imaging procedure | During the procedure
  Length of acquisition time from the first to the last images
Secondary effects | From Procedure until 2 days after
  Number of participant developing any secondary effects
Failure of pentobarbital sedation in children older than 5 years | During the procedure
  Comparison of the rate of failure of pentobarbital sedation in children older than 5 years compared to those younger.
Failure of pentobarbital sedation in children with a behavioral disorder | During the procedure
  Comparison of the rate of failure of pentobarbital sedation in children with a behavioral disorder compared to those without
Failure of pentobarbital sedation in children under chronic antiepileptic treatment | During the procedure
  Comparison of the rate of failure of pentobarbital sedation in children under chronic antiepileptic treatment compared to those without

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Ropars, MD, Study Director — Brest University Hospital in France
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No